CLINICAL TRIAL: NCT02940184
Title: Vagal Mechanisms Mediating the Effects of Glucagon-Like Peptide 1 (GLP-1) on the Endocrine Pancreas - the Entero-endocrine Axis.
Brief Title: GLP-1 Signaling in Truncally Vagotomized Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Simon Veedfald, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UC/RH-vago-GLP-1
Record Dates: First submitted 2016-04-07; First posted 2016-10-20 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Physiology
Keywords: Physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteral fructose with DPP-4 inhibition (Experimental): Enteral fructose + DPP-4 inhibition (sitagliptin)
  After DPP4 inhibition using Tablet Sitagliptin 100mg on the evening before and on the morning of experimentation enteral fructose is given via an intestinal tube (intrajejunal) to either truncally vagotomised and control individuals.
  Interventions: Drug: Tablet Sitagliptin 100mg (evening before and morning of experiments); Other: Intestinal Fructose administration
- Enteral fructose without DPP-4 inhibition (Experimental): Enteral fructose without DPP-4 inhibition (sitagliptin) After DPP4 inhibition using Tablet Sitagliptin 100mg on the evening before and on the morning of experimentation enteral fructose is given via an intestinal tube (intrajejunal) to either truncally vagotomised and control individuals.
  Interventions: Other: Intestinal Fructose administration

INTERVENTIONS:
Drug: Tablet Sitagliptin 100mg (evening before and morning of experiments) — On one of two experiment days participants will have Dipeptidyl peptidase 4 activity inhibited using a DPP-4 inhibitor (Sitagliptin).
  Arms: Enteral fructose with DPP-4 inhibition
Other: Intestinal Fructose administration — On both experimental days fructose (35g dissolved in water, total volume 100mL) will be administered via an intrajejunal tube

SUMMARY:
Investigation of the importance of vagal signaling for the glucohomeostatic effects of GLP-1. The study will include physiological studies of truncally vagotomized participants and matched controls.

ELIGIBILITY:
Truncally vagotomized individuals:

Inclusion Criteria:

* Normal fasting plasma glucose
* Normal haemoglobin concentration
* Cardiaresection with a pyloroplasty
* Informed consent

Exclusion Criteria:

* Diabetes mellitus
* Disposition for diabetes mellitus
* Intestinal disease (apart from cardia resection+pyloroplasty)
* Disposition of inflammatory bowel disease
* Intestinal resection (apart from cardia resection+pyloroplasty)
* Body mass index (BMI) > 27,5 kg/m2
* Tobacco use
* Nephropathy (se-creatinine> 130 µM and/or albuminuria)
* Liver disease (ALAT and/or ASAT >2 × refference value)
* known heart condition
* medicinal use, that may not be paused for 12 hours
* Obstipation
* swallowing difficulties
* previous problems with intestinal tube placement
* Latex allergy
* Fructose malabsorption
* Known diseases in the pharynx
* Previous facial or cranial fractures
* Sinusitis
* Bleeding diathesis

Matched controls:

Inclusion Criteria:

* Normal fasting plasma glucose
* Normal haemoglobin concentration
* Informed consent

Exclusion Criteria:

* Cardiaresection with a pyloroplasty
* Diabetes mellitus
* Disposition for diabetes mellitus
* Intestinal disease (apart from cardia resection+pyloroplasty)
* Disposition of inflammatory bowel disease
* Intestinal resection tarmresektion (apart from cardia resection+pyloroplasty)
* Body mass index (BMI) > 27,5 kg/m2
* Tobacco use
* Nephropathy (se-creatinine> 130 µM and/or albuminuria)
* Liver disease (ALAT and/or ASAT >2 × refference value)
* known heart condition
* medicinal use, that may not be paused for 12 hours
* Obstipation
* swallowing difficulties
* previous problems with intestinal tube placement
* Latex allergy
* Fructose malabsorption
* Known diseases in the pharynx
* Previous facial or cranial fractures
* Sinusitis
* Bleeding diathesis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Insulin secretion | up to 4 hours
  Evaluated by c-peptide and insulin levels - Plasma collected up to 4 hours will be analyzed for peptide hormones

SECONDARY OUTCOMES:
Glucagon secretion | 4 hours
  Plasma collected over 4 hours will be analyzed for peptide hormones
Glucose levels | 4 hours
  Plasma collected over 4 hours will be analyzed for glucose
Pancreatic Polypeptide levels | 4 hours
  Plasma collected over 4 hours will be analyzed for peptide hormones
GIP secretion | 4 hours
  Plasma collected over 4 hours will be analyzed for peptide hormones

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery C, Rigshospitalet, Copenhagen, Denmark